CLINICAL TRIAL: NCT00109200
Title: A Continued Access Protocol to Provide Xolair® (Omalizumab) to Subjects With Severe Allergic Asthma Who Have Received Xolair Treatment in a Previous Investigational Study
Brief Title: A Continued Access Protocol to Provide Xolair to Patients With Severe Allergic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: Q2736g
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Allergic Asthma; Severe Allergic Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: Xolair (omalizumab)

SUMMARY:
This is a continued access protocol to provide subjects who have completed Genentech, Inc. Study Q2143g, Q2195g, or Q2461g or Novartis Pharmaceuticals Corporation Study CIGE025 0010E1 with continued Xolair treatment. Subject eligibility will be based on disease severity and asthma deterioration upon withdrawal of Xolair treatment. Subjects whose last Xolair dose was <9 months prior to screening visit will continue with the same Xolair dosing regimen that they received in the previous Genentech or Novartis clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of Genentech Study Q2143g, Q2195g, or Q2461g or Novartis Study CIGE025 0010E1
* Signed informed consent document (in the case of a minor, consent must be given by the child's parent or legally authorized representative)
* Females of childbearing potential must, in the opinion of the investigator, be using an effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
* Severe asthma as demonstrated by at least one of the following: *History of prior intubation for allergic asthma; *History of prior admission to an intensive care unit/pediatric ICU for asthma; *History of one or more hospitalizations, emergency room (ER) visits, or unscheduled office visits for asthma in the 12 months prior to first Xolair treatment; *More than 20 days missed from school/work because of allergic asthma in the 12 months prior to initiation of Xolair treatment
* Deterioration of asthma upon withdrawal of Xolair as demonstrated by meeting at least one of the following: *Worsening of pulmonary function tests (FEV1 <80% predicted for height, age, and sex) and activity levels while off Xolair treatment; *Worsening of asthma exacerbations defined as doubling of inhaled steroid dose, increase in dose of oral steroids, or initiation of oral, intravenous, intramuscular, or subcutaneous (SC) steroids while off Xolair treatment; *Increased use of rescue medications while off Xolair treatment; *ER visits or unscheduled office visits for asthma that may or may not result in hospitalization while off Xolair treatment

Exclusion Criteria:

* Pregnancy or lactation
* Significant systemic disease (e.g., hematologic, renal, hepatic, coronary heart, endocrine, gastrointestinal disease, other cardiovascular diseases, or infection) within the previous 3 months
* History of neoplasia (including basal cell carcinoma)
* Any systemic condition requiring regular administration of an immunoglobulin
* Known hypersensitivity to any ingredients of Xolair, including excipients (sucrose, histidine, polysorbate 20)
* Current treatment with warfarin (Coumadin(R)), immunomodulatory therapy (e.g., methotrexate, gold, cyclosporine), or antiplatelet therapy
* Current participation in a study using an investigational new drug other than Xolair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-05; Study Completion 2003-09 (Actual)